CLINICAL TRIAL: NCT02259608
Title: Training of Innate Immunity by Vaccination With γ-irradiated BCG
Brief Title: γ-irradiated BCG to Train Innate Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL45427.091.13; 2013/319 (Other: CMO Arnhem Nijmegen)
Record Dates: First submitted 2014-09-26; First posted 2014-10-08 (Estimated); Results first posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-01

CONDITIONS: Innate Immune Response
Keywords: Trained innate immunity; Heterologous effects of BCG on immunity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BCG vaccine SSI (Experimental): Healthy volunteers are vaccinated with yBCG. Blood will be drawn before and at several timepoints after vaccination. Cytokine production before vaccination will be used as reference to compare later timepoints with.
  Interventions: Biological: BCG vaccine SSI

INTERVENTIONS:
Biological: BCG vaccine SSI — BCG vaccination
  Other Names: J07AN01

SUMMARY:
Rationale: The live attenuated Bacillus Calmette-Guerin (BCG) vaccine protects against extrapulmonary infection with Mycobacterium tuberculosis and leprosy. It has been shown that vaccination with BCG also leads to nonspecific protective effects, e.g. reduced infant mortality as a result of less severe infections, stimulation of the immune system in patients with bladder cancer and higher cytokine production upon restimulation of macrophages with non-related infectious pathogens in vitro. However, because the live attenuated BCG vaccine cannot be used in immune compromised hosts, the investigators would like to determine whether similar protective non-specific effects can be induced by γ-irradiated BCG.

Objective: To determine whether vaccination with γ-irradiated BCG results in a higher cytokine response by monocytes upon restimulation in vitro with infectious pathogens, compared to monocytes before the vaccination.

Study design: Explorative intervention trial. Study population: Healthy volunteers, 18 - 55 years old. Intervention: Healthy volunteers will be vaccinated with γ-irradiated BCG vaccine.

Main study parameters/endpoints: Blood will be drawn before and at two different time points after vaccination with BCG to perform restimulation of isolated cells in vitro and compare cytokine production.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is no known direct benefit for the volunteers to participate in the trial. The risks are negligible. BCG vaccination can cause pain and scarring at the site of injection, just as fever and headache. Local hematoma formation can occur at the site of the blood drawing. This will be minimized by the blood collection by experienced persons.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   The live attenuated Bacillus Calmette-Guerin (BCG) vaccine protects against extrapulmonary infection with Mycobacterium tuberculosis and against leprosy [1, 2]. It has been shown that vaccination with BCG also leads to non-specific protective effects: early administration of BCG vaccination could lead to reduced child mortality, mainly as a result of reduced neonatal sepsis, respiratory infection, and fever. [3-5] Furthermore, BCG has also been used in patients with bladder cancer, to induce an improved reaction of the immune system, which prevents tumor progression and dead. [6] Recently, it was shown that BCG vaccination can induce epigenetic changes in human monocytes, which result in higher pro-inflammatory cytokines response upon restimulation with non-related pathogens in vitro. [7] The observed effects are proposed to be due to modulation of the human innate immune system, in a process called 'trained immunity'. Upon stimulation with a pathogen, the innate immune system becomes primed and is able to react faster and more efficient to a secondary (and non-related) stimulus. [7, 8]

   Considering these beneficial effects of BCG on innate host defense, it is reasonable to hypothesize that it would be helpful to generate a 'trained immunity status' in hosts defective in T- and B-cell immunity, as they are more vulnerable to infections. However, because of their immune compromised status, these patients cannot be vaccinated with live attenuated vaccines (e.g. BCG). [9] Vaccination with y-irradiated BCG would be possible, but it is not known whether the γ-irradiated vaccine has the same protective non-specific effects on innate host defense. In recent in-vitro experiments, the investigators have demonstrated that y-irradiated BCG can train monocytes in vitro (not published). Therefore, the aim of this study is to determine whether γ-irradiated BCG is able to train the human innate immune system of healthy volunteers in-vivo, just as shown before with the live attenuated BCG vaccine [7].
2. OBJECTIVES

   Primary Objective: To determine whether γ-irradiated BCG can train the innate immune system in vivo, by comparing cytokine production upon ex-vivo restimulation with pathogens before, 2 weeks and 3 months after vaccination with y-irradiated BCG.
3. STUDY DESIGN

   An explorative intervention study with a duration of three months will be performed. 15 Healthy volunteers will be recruited to receive a vaccination with γ-irradiated BCG. After informed consent, 40ml of blood will be drawn before vaccination and at 2 weeks and 3 months post-vaccination.
4. STUDY POPULATION 4.1 Population Healthy volunteers, 18 - 55 yr old. 4.2 Inclusion criteria The subjects must be healthy adults, aged 18 - 55 years old. 4.3 Exclusion criteria Subjects are excluded when they are from tuberculosis endemic countries, if they have been in contact with tuberculosis patients or if they already have been vaccinated with BCG. The subjects are excluded from the study if they suffer for any disease, including intercurrent infections. Subjects are not allowed to use any medication except oral anticonceptive agents.

   4.4 Sample size calculation This is an explorative trial, for which sample size calculation is not possible.
5. TREATMENT OF SUBJECTS 5.1 Investigational product/treatment Subjects will be vaccinated with a y-irradiated BCG vaccine (BCG-Vaccin SSI [Nederlands Vaccin Instituut]), which is purchased from Radboud Apotheek B.V.

   γ-Irradiation of the BCG vaccine will be performed by Synergy Health Ede B.V., Ede, The Netherlands (registered by the Dutch Ministry of Economic Affairs). The BCG vaccine was radiated in the original packaging with an average dose of 32.2kGy in a JS6500 Tote Box Irradiator. This dose is based on an in the literature accepted minimal dose of 25kGy, which has been proven to be sufficient to kill M. tuberculosis [10, 11] . After irradiation the vaccine will be returned unopened in the original packaging. During the irradiation a dosimeter is included, so each irradiated batch will come along with a certificate with the exact irradiation dose used.

   5.2 Use of co-intervention Subjects are not allowed to use any medication, except for oral anticonception.
6. INVESTIGATIONAL PRODUCT 6.1 Name and description of investigational product(s) y-Irradiated BCG vaccine (BCG-Vaccin SSI [Nederlands Vaccin Instituut]) Danish strain 1331.

   6.2 Summary of findings from non-clinical studies The efficacy of killing by γ-irradiating of the BCG vaccine was verified by culturing the y-irradiated BCG in special tuberculosis culture medium. No growth was detected after six weeks.

   6.3 Summary of findings from clinical studies A related study with a comparable study setup, in which 20 healthy volunteers were vaccinated with live attenuated BCG vaccine has already been accomplished. [7] The investigators study will use the same study protocol. The only difference is that instead of the live attenuated BCG vaccine a y-irradiated BCG vaccine will be used.

   6.4 Summary of known and potential risks and benefits There are no clear benefits for the volunteers. Potential risks are very small, as BCG is considered a safe vaccine. BCG vaccination can cause pain and scarring at the site of injection just as fever and headache, and very sporadic occurring side effects as syncope, convulsions and allergic reaction. Local hematoma formation can occur at the site of the blood drawing.

   6.5 Description and justification of route of administration and dosage Administer at the upper arm slowly, in about 10 seconds, intracutaneous 0.1ml of the suspended vaccine, which accounts for 0.075mg of Mycobacterium bovis.
7. METHODS 7.1 Study parameters/endpoints Before the vaccination and at two different time points after vaccination with γ-irradiated BCG (2 weeks and 3 months) blood will be drawn, from which PBMCs will be isolated by density centrifugation over Ficoll-Paque. Monocytes will be restimulated ex-vivo with different pathogens (M. tuberculosis (1µg/ml), S. aureus, C. albicans (both 1 x 10^6 microorganisms/ml), and E. coli LPS (10ng/ml). Cytokine production will be assessed after 24h (TNFa, IL 1b and IL-6), 48h (IFN, IL-10) and 7 days (IL-17, IL-22) stimulation, and compared with cytokine production before vaccination.

7.2 Study procedures Subjects will be vaccinated with y-irradiated BCG vaccine. Before and twice after vaccination, 40ml of blood will be drawn.

7.3 Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences.

7.4 Replacement of individual subjects after withdrawal Each withdrawn subject will be replaced, in order that in total 15 subjects will complete the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must be healthy adults, aged 18 - 55 years old

Exclusion Criteria:

* Subjects are excluded when they are from tuberculosis endemic countries, if they have been in contact with tuberculosis patients or if they have been earlier vaccinated with BCG.
* The subjects are excluded from the study if they suffer for any disease, including intercurrent infections.
* Subjects are not allowed to use any medication except oral anticonceptive agents.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCG Vaccine SSI
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- yBCG: 15 healthy volunteers that receive yBCG at baseline. There is no control group included in this trial.
Arm/Group | yBCG
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 23 [20 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Healthy [Number; unit: participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: Cytokine Production Measured by ELISA Compared to Baseline
Description: Comparing tnfa production of PBMCs after 24h stimulation with candida before and 3 months after yBCG vaccination.
  Baseline is set as 1.
Time Frame: 0 weeks and 3 months
Population: Ex-vivo cytokine production by PBMCs upon stimulation with several pathogens
Measure: Mean (Full Range); unit: ratio
Arm/Group | BCG Vaccine SSI
Number analyzed (Participants) | 15
ratio | 1.2 [0.5 to 2.2]

2. Secondary Outcome: Cytokine Production Measured by ELISA Compared to Baseline
Description: Ex-vivo cytokine production by PBMCs upon stimulation with several pathogens
Time Frame: 0 weeks and 2 weeks
Measure: Mean (Full Range); unit: ratio
Arm/Group | BCG Vaccine SSI
Number analyzed (Participants) | 15
ratio | 1.4 [0.6 to 3.4]

ADVERSE EVENTS:
Arm/Group | BCG Vaccine SSI
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCG Vaccine SSI (N=15)
Local reaction to BCG vaccin (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes